CLINICAL TRIAL: NCT00363363
Title: Identifying Determinants and Optimizing Rehabilitation of Physical Activity for Children After the Fontan Procedure
Brief Title: Physical Activity in Fontan Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000008413
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Heart Defects, Congenital
Keywords: Pediatrics; Fontan Procedure; Physical Activity; Physical Fitness; Congenital Heart Defects; exercise rehabilitation
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Physical Activity
- 2 (Active Comparator)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Physical Activity — Children in this arm of the study will be provided with specific activities to be completed on most days of the week. The selected activities will be based on the child's interests and results of the baseline measures of health-related PA, MVPA and gross motor skill. The resources and facilities available to the family and season of the year will also influence the choice of activities. The frequency and duration of the required activities will be gradually increased until the child's baseline MVPA has been increased by a minimum of 30 minutes per day, most days of the week. Once that increase is achieved, the activities will be modified to maintain and reinforce the higher PA level.
  Arms: 1
Behavioral: Education — Children in this arm of the study will be provided with puzzles, stories and games to be completed each week. The selected activities will be based on the child's interests and designed to increase the child's knowledge of activity options, perceptions of activity benefits, self-confidence for activity participation and motivation for daily activity. The activities introduced will vary with the resources available to the family and the season of the year, and will include information about healthy eating, injury prevention, and healthy lifestyle options.
  Arms: 2

SUMMARY:
The purpose of this study is to determine which is the most effective intervention for increasing lifestyle physical activity in Fontan patients: an education (stage of change) intervention or a physical activity (mastery experience) intervention.

DETAILED DESCRIPTION:
Over 100,000 Canadian children are living with congenital heart defects and approximately 1.5% of them have a univentricular heart. The Fontan procedure allows children with functionally univentricular hearts to live relatively normal lives. However, the cardiopulmonary physiology remains abnormal and chronic complications, including myocardial dysfunction, arrhythmias, pathway abnormalities, hepatic dysfunction, obstruction of the ventricular outflow tract or pulmonary veins, and pulmonary arteriovenous malformations may significantly reduce maximal exercise capacity and quality of life. Quality of life and life-long heart health are, therefore, critically important for Fontan patients as their survival depends on the continued functioning of an already sub-normal cardiopulmonary physiology.

ELIGIBILITY:
Inclusion Criteria:

* have undergone a successful Fontan procedure prior to 5 years of age
* 6 to 10 years of age at the start of the study
* sufficient cardiopulmonary function (based on pulmonary function tests prior to the standardized cardiorespiratory exercise test) for safe participation in moderate to vigorous physical activity

Exclusion Criteria:

* disabilities or medical conditions that may influence physical activity participation.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in the child's moderate-to-vigorous physical activity participation | From baseline to end of treatment (12 months) and follow up (6-12 months post-treatment)

SECONDARY OUTCOMES:
Increase in health-related physical fitness | From baseline to end of treatment (12 months) and follow up (6-12 months post-treatment)
Achievement of age-appropriate gross motor skills | From baseline to end of treatment (12 months) and follow up (6-12 months post-treatment)
Change in the parents' and child's perceptions of physical activity importance, value, appropriateness and competence | From baseline to end of treatment (12 months) and follow up (6-12 months post-treatment)
Compliance with the intervention | From baseline to end of treatment (12 months) and follow up (6-12 months post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada